CLINICAL TRIAL: NCT00437762
Title: Effectiveness of Botulinum Toxin A Injection for the Treatment of Lateral Epicondylitis Unrelieved by Usual Medical Cares : A Double Blind Randomized Controlled Trial Versus Placebo
Brief Title: Effectiveness of Botulinum Toxin Injection in the Tennis Elbow Treatment
Acronym: TBA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2005/08
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Tennis Elbow
Keywords: Lateral epicondylitis, tennis elbow, treatment
MeSH Terms: conditions — Tennis Elbow | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Botulinum Toxin A Injection
  Interventions: Drug: Botulinum Toxin A Injection
- 2 (Placebo Comparator): Placebo injection
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Botulinum Toxin A Injection — Botulinum Toxin A Injection
  Arms: 1
Drug: Placebo injection — Placebo Injection
  Arms: 2

SUMMARY:
Some studies valued the effectiveness of botulinum toxin. Results are contradictory and we need more studies. The purpose of the study is to compare the effectiveness of botulinum toxin injection with placebo in the treatment of tennis elbow unrelieved by usual medical care performed during 6 months. Method : It is a double blind randomized controlled trial. Principal criteria of assessment is Pain intensity three months after injection.

DETAILED DESCRIPTION:
* Principal Objective : The first aim of the study is to value the effectiveness of botulinum toxin injection in the treatment of tennis elbow unrelieved by usual medical care performed during 6 months..
* Secondary Objective : The second aim of this study is to document the tennis elbow history by a one year following after initial injection
* Study design : It is a double blind randomized controlled trial. Principal criteria of assessment is Pain intensity three months after injection.
* Inclusion criteria : tennis elbow during more than 6 months ; signature of consent
* Exclusion criteria : Non inclusion criteria : less than 18 years old ; osteoarthritis elbow, referred cervical pain, fibromyalgia, pregnancy, myasthenia, polymyositis, SLA, anticoagulant treatment, aminosides ; diabetes, alcoholism
* Study plan: randomized parallel groups
* Number of subjects : 60

ELIGIBILITY:
Inclusion Criteria:

* Tennis elbow during more than 6 months
* Signature of consent

Exclusion Criteria:

* Less than 18 years old
* Osteoarthritis elbow
* Referred cervical pain
* Fibromyalgia
* Pregnancy
* Myasthenia
* Polymyositis
* SLA
* Anticoagulant treatment
* Aminosides
* Diabetes
* Alcoholism
* Previous botulinum toxin A injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Principal criteria of assessment is pain intensity three months after injection. | at 3 month

SECONDARY OUTCOMES:
pain intensity | to day 30, 90,180, 365
Number of painful days | to day 30, 90,180, 365
Number of associated treatments. | to day 30, 90,180, 365
Free pain grip strength | to day 30, 90,180, 365
Rate of recidivism after initial relief | to day 30, 90,180, 365

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu DE SEZE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Unité de médecine orthopédique- Hôpital Pellegrin RDC aile 2., Bordeaux, France